CLINICAL TRIAL: NCT00668525
Title: A Double-blind, Fixed-dose Study of Escitalopram in Adult Patients With Major Depressive Disorder
Brief Title: Escitalopram in Adult Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Carl Gommoll, Study Director, Forest Laboratories
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCT-MD-49
Record Dates: First submitted 2008-04-28; First posted 2008-04-29 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; Escitalopram
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): Escitalopram low dose
  Interventions: Drug: Escitalopram
- 3 (Experimental): Escitalopram high dose
  Interventions: Drug: Escitalopram
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram low dose, oral administration, once daily dosing for 8 weeks.
  Arms: 2
Drug: Placebo — Placebo, oral administration, once daily dosing for 8 weeks
  Arms: 1
Drug: Escitalopram — Escitalopram high dose, oral administration, once daily dosing for 8 weeks
  Arms: 3

SUMMARY:
This is a short-term study to evaluate the efficacy, safety, and tolerability of escitalopram in adult patients (18 to 65 years of age) with moderate to severe depression. Patients completing the study may be eligible to enter a long-term open-label extension study with escitalopram.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR) diagnostic criteria for Major Depressive Disorder.
* The patient's current depressive episode must be at least 8 weeks in duration.

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not practicing a reliable method of birth control.
* Patients with a history of meeting DSM-IV-TR criteria for: a. any manic or hypomanic episode; b. schizophrenia or any other psychotic disorder; c. obsessive-compulsive disorder.
* Patients who are considered a suicide risk
* Patients with a history of seizures (including seizure disorder), stroke, significant head injury, central nervous system tumors, or any other condition that predisposes patients to a risk for seizure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Laboratories
Locations (42):
- United States (42):
  - Forest Investigative Site, Phoenix, Arizona
  - Forest Investigative Site, Arcadia, California
  - Forest Investigative Site, Encino, California
  - Forest Investigative Site, Garden Grove, California
  - Forest Investigative Site, Irvine, California
  - Forest Investigative Site, Los Alamitos, California
  - Forest Investigative Site, Denver, Colorado
  - Forest Investigative Site, Washington D.C., District of Columbia
  - Forest Investigative Site, Bradenton, Florida
  - Forest Investigative Site, Jacksonville, Florida
  - Forest Investigative Site, Orlando, Florida
  - Forest Investigative Site, West Palm Beach, Florida
  - Forest Investigative Site, Atlanta, Georgia
  - Forest Investigative Site, Newton, Kansas
  - Forest Investigative Site, Overland, Kansas
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site, Glen Burnie, Maryland
  - Forest Investigative Site, Rockville, Maryland
  - Forest Investigative Site, Okemos, Michigan
  - Forest Investigative Site, St Louis, Missouri
  - Forest Investigative Site, Omaha, Nebraska
  - Forest Investigative Site, Cherry Hill, New Jersey
  - Forest Investigative Site, Clementon, New Jersey
  - Forest Investigative Site, Brooklyn, New York
  - Forest Investigative Site, New York, New York
  - Forest Investigative Site, Staten Island, New York
  - Forest Investigative Site, The Bronx, New York
  - Forest Investigative Site, Canton, Ohio
  - Forest Investigative Site, Dayton, Ohio
  - Forest Investigative Site, Portland, Oregon
  - Forest Investigative Site, Media, Pennsylvania
  - Forest Investigative Site, Philadelphia, Pennsylvania
  - Forest Investigative Site, Charleston, South Carolina
  - Forest Investigative Site, Memphis, Tennessee
  - Forest Investigative Site, Austin, Texas
  - Forest Investigative Site, Houston, Texas
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Salt Lake City, Utah
  - Forest Investigative Site, Woodstock, Vermont
  - Forest Investigative Site, Richmond, Virginia
  - Forest Investigative Site, Bellevue, Washington
  - Forest Investigative Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 4/30/08 through 12/19/08 with last patient last visit on 2/24/09 at 45 centers in the US.
Pre-assignment Details: A one-week single-blind placebo period was completed prior to randomization. Patients were then randomized in a 3:3:2 ratio to either escitalopram low dose, escitalopram high dose or placebo.
Groups:
- Escitalopram Low Dose: Escitalopram low dose, administered orally (QD [once a day]) for 8 weeks of stable dose treatment phase. The Overall Number of Baseline Participants is based on the Safety population.
- Escitalopram High Dose: Escitalopram high dose, administered orally (QD [once a day]) for 8 weeks of stable dose treatment phase. The Overall Number of Baseline Participants is based on the Safety population.
- Placebo: Placebo, administered orally (QD [once a day]) for 8 weeks of stable dose treatment phase. The Overall Number of Baseline Participants is based on the Safety population.
Period: Overall Study
Arm/Group | Escitalopram Low Dose | Escitalopram High Dose | Placebo
Started | 325 (The number of patients started are based on the Randomized Population.) | 332 (The number of patients started are based on the Randomized Population.) | 220 (The number of patients started are based on the Randomized Population.)
Completed | 248 (The number of patients completed are based on the Randomized Population.) | 239 (The number of patients completed are based on the Randomized Population.) | 167 (The number of patients completed are based on the Randomized Population.)
Not Completed | 77 | 93 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram Low Dose | Escitalopram High Dose | Placebo | Total
Number analyzed (Participants) | 322 | 324 | 218 | 864
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 322 | 324 | 218 | 864
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.3) | 40.4 (11.9) | 42.3 (12.7) | 41.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 222 | 137 | 564
  Male | 117 | 102 | 81 | 300
Region of Enrollment [Number; unit: participants]
  United States | 322 | 324 | 218 | 864

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Montgomery Asberg Depression Rating Scale (MADRS) at 8 Weeks.
Description: The MADRS is a 10-item clinician-rated scale that was used to assess depressive symptomatology over the patient's prior week. Patients were rated on 10 items designed to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest. Each item was scored on a 7-point Likert scale; a score of 0 indicated the absence of symptoms, and a score of 6 indicated symptoms of maximum severity. The total score range is 0 to 60 (higher score indicates a greater severity of symptoms).
Time Frame: Change from baseline in MADRS total score at week 8
Population: The analysis was performed on the intent to treat population based on the LOCF approach using an ANCOVA model with treatment group and study center as factors and the baseline MADRS total score as a covariate.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Escitalopram Low Dose | Escitalopram High Dose | Placebo
Number analyzed (Participants) | 319 | 318 | 215
Units on a scale | -12.8 (0.6) [-4.6 to -1.2] | -13.4 (0.6) [-1.9 to 1.1] | -10.1 (0.7) [-5.0 to -1.6]

2. Secondary Outcome: Change From Baseline in Hamiltion Rating Scale for Depression (HAM-D) at Week 8
Description: The HAMD is a clinician-rated 24-item scale was used to rate the patient's depressive state. It was also used to identify obsessive-compulsive, genital, and somatic symptoms, as well as diurnal variation in the presence of symptoms. Each item was scored on a 3, 4 or 5-point Likert scale. A score of 0 indicated the absence of symptoms, and a score of 2, 3 or 4 indicated symptoms of maximum severity. The total score range is 0 to 74 (higher score indicates a greater depressive state).
Time Frame: Change from baseline in HAM-D at week 8
Population: The analysis was performed on the intent to treat population based on the LOCF approach using an ANCOVA model with treatment group and study center as factors and the baseline HAMD total score as a covariate.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Escitalopram Low Dose | Escitalopram High Dose | Placebo
Number analyzed (Participants) | 319 | 318 | 215
Units on a scale | -11.5 (0.5) | -11.6 (0.6) | -8.5 (0.6)

ADVERSE EVENTS:
Time Frame: 10 months.
Arm/Group | Escitalopram Low Dose | Escitalopram High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 3/322 | 7/324 | 4/218
Other Adverse Events (participants affected / at risk) | 146/322 | 160/324 | 74/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram Low Dose (N=322) | Escitalopram High Dose (N=324) | Placebo (N=218)
Chest Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple Sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram Low Dose (N=322) | Escitalopram High Dose (N=324) | Placebo (N=218)
Headache (Nervous system disorders) | 52 | 45 | 31
Nausea (Gastrointestinal disorders) | 41 | 37 | 16
Diarrhea (Gastrointestinal disorders) | 30 | 35 | 14
Insomnia (Psychiatric disorders) | 19 | 34 | 7
Dry mouth (Gastrointestinal disorders) | 23 | 28 | 7
Somnolence (Nervous system disorders) | 17 | 26 | 4
Fatigue (General disorders) | 18 | 20 | 4
Dizziness (Nervous system disorders) | 15 | 14 | 12
Nasopharyngitis (Infections and infestations) | 6 | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 90 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential info. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in pub. On sponsor's request, PI shall delay submission for any pub while sponsor files patent apps. If trial is multi-center, PI agrees that first publication shall be a multi-center pub.